CLINICAL TRIAL: NCT03247114
Title: Functional Magnetic Resonance Imaging of Human Hypothalamic Responses to Glucose, Fructose, Sucrose and Sucralose
Brief Title: fMRI of Hypothalamic Responses to Glucose, Fructose, Sucrose and Sucralose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1930
Record Dates: First submitted 2017-08-07; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Healthy
MeSH Terms: interventions — Water; Glucose; Fructose; Sucrose; trichlorosucrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Water-glucose-sucralose-fructose-sucrose (Experimental): First plain water, then glucose, then sucralose, then fructose and then sucrose
  Interventions: Other: Water; Other: Glucose; Other: Fructose; Other: Sucrose; Other: Sucralose
- water-sucralose-glucose-sucrose-fructose (Experimental): First plain water, then sucralose, then glucose, then sucrose and then fructose
  Interventions: Other: Water; Other: Glucose; Other: Fructose; Other: Sucrose; Other: Sucralose
- Glucose-water-fructose-sucralose-sucrose (Experimental): First glucose, then plain water, then fructose, then sucralose and then sucrose
  Interventions: Other: Water; Other: Glucose; Other: Fructose; Other: Sucrose; Other: Sucralose
- Glucose-fructose-water-sucrose-sucralose (Experimental): First glucose, then fructose, then plain water, then sucrose and then sucralose
  Interventions: Other: Water; Other: Glucose; Other: Fructose; Other: Sucrose; Other: Sucralose
- Fructose-glucose-sucrose-water-sucralose (Experimental): First fructose, then glucose, then sucrose, then plain water and then sucralose
  Interventions: Other: Water; Other: Glucose; Other: Fructose; Other: Sucrose; Other: Sucralose
- Fructose-sucrose-glucose-sucralose-water (Experimental): First fructose, then sucrose, then glucose, then sucralose and then plain water
  Interventions: Other: Water; Other: Glucose; Other: Fructose; Other: Sucrose; Other: Sucralose
- Sucrose-fructose-sucralose-glucose-water (Experimental): First sucrose, then fructose, then sucralose, then glucose and then plain water
  Interventions: Other: Water; Other: Glucose; Other: Fructose; Other: Sucrose; Other: Sucralose
- Sucrose-sucralose-fructose-water-glucose (Experimental): First sucrose, then sucralose, then fructose, then plain water and then glucose
  Interventions: Other: Water; Other: Glucose; Other: Fructose; Other: Sucrose; Other: Sucralose
- Sucralose-water-sucrose-glucose-fructose (Experimental): First sucralose, then plain water, then sucrose, then glucose and then fructose
  Interventions: Other: Water; Other: Glucose; Other: Fructose; Other: Sucrose; Other: Sucralose
- Sucralose-sucrose-water-fructose-glucose (Experimental): First sucralose, then sucrose, then plain water, then fructose and then glucose
  Interventions: Other: Water; Other: Glucose; Other: Fructose; Other: Sucrose; Other: Sucralose

INTERVENTIONS:
Other: Water — Water, 300 ml at room temperature
Other: Glucose — Glucose, 50 grams in 300 ml water at room temperature
Other: Fructose — Fructose, 50 grams in 300 ml water at room temperature
Other: Sucrose — Sucrose, 50 grams in 300 ml water at room temperature
Other: Sucralose — Sucralose, 0.33 grams in 300 ml water at room temperature

SUMMARY:
The study will consist of five occasions with one week in between. BOLD signal intensity of the hypothalamus will be measured using fMRI. Measurements will be done before and after drinking 300 ml plain water (reference) or water to which different sweeteners will be added.

DETAILED DESCRIPTION:
The hypothalamus is known to be important for control of feeding behaviour as well as the regulation of temperature. Functional magnetic resonance imaging (fMRI) is a non-invasive method, which detects transient haemodynamic changes in the brain, using blood oxygen level dependent (BOLD) signal differences.

In order to investigate the role of hypothalamic neural activity in response to different sweeteners, fMRI will be performed before, during and after ingestion of 300 ml plain water or 300 ml water containing 50 g glucose, 50 g fructose, 50 g sucrose or 0.33 g sucralose (high intensity sweetener not providing energy). All beverages will be consumed at 22 °C.

The study uses a randomized cross-over design in 16 healthy male subjects with a normal body weight. There will be an interval of at least one week between the five occasions.

Blood Oxygen Level Dependent signal intensity of the hypothalamus will be continuously measured for 21 minutes (5 minutes baseline, 4 minutes during drinking and 12 minutes after drinking).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between 18 and 25 years
* BMI between 20 and 24 kg/m2
* Length between 170 and 190 centimetres

Exclusion Criteria:

* Diabetes or history of other disturbances of glucose metabolism (eg impaired glucose tolerance, hypoglycaemia).
* Any genetic or psychiatric disease (e.g. fragile X syndrome, major depression) affecting brain
* Any significant chronic disease
* Renal or hepatic disease
* Recent weight changes or attempts to lose weight (> 3 kg weight gain or loss, within the last 3 months)
* Smoking (current or last 6 months)
* Alcohol consumption of more than 21 units per week or use of recreational drugs at present or in the last year
* Recent blood donation (within the last 2 months)
* Recent participation in other biomedical research projects (within the last 3 months), participation in 3 or more biomedical research projects in one year
* Contra-indication to MRI scanning:

  * Claustrophobia
  * Pacemakers and defibrillators
  * Nerve stimulators
  * Intracranial clips
  * Intraorbital or intraocular metallic fragments
  * Cochlear implants
  * Ferromagnetic implants

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02-22 (Actual); Primary Completion 2015-05-22 (Actual); Study Completion 2015-05-22 (Actual)

PRIMARY OUTCOMES:
Hypothalamic function in response to glucose, fructose, sucrose, and sucralose | Change from baseline (measured during 5 minutes before start of dinking) to post consumption (measured during 12 minutes after drinking). Drinking took 4 minutes.
  fMRI will be performed before and after ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen van der Grond, Dr, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leids Universitair Medisch Centrum, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Opstal AM, Hafkemeijer A, van den Berg-Huysmans AA, Hoeksma M, Blonk C, Pijl H, Rombouts SARB, van der Grond J. Brain activity and connectivity changes in response to glucose ingestion. Nutr Neurosci. 2020 Feb;23(2):110-117. doi: 10.1080/1028415X.2018.1477538. Epub 2018 May 27. PMID 29806553